CLINICAL TRIAL: NCT06493968
Title: Role of Uterotonics in Reducing Intraoperative Blood Loss in Patients With Placenta Accrete Spectrum Disorders Undergoing Cesarean Hysterectomy
Brief Title: Role of Uterotonics in Reducing Intraoperative Blood Loss in Patients With PASD Undergoing Cesarean Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer of obgyn Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Uterotonics in PASD
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): Patients will be given uterotonics
  Interventions: Drug: oxytocin
- Group (B) (Placebo Comparator): Patients will not be given uterotonics
  Interventions: Other: placebo

INTERVENTIONS:
Drug: oxytocin — Uterotonics will be given in the form of an IV bolus of 10 units of oxytocin immediately with the uterine incision
  Arms: Group (A)
Other: placebo — IV bolus of normal saline immediately with the uterine incision
  Arms: Group (B)

SUMMARY:
Objectives: To evaluate the effect of oxytocin in reducing intraoperative blood loss in patients with PAS disorders planned for cesarean hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy of singleton living fetus
* Previous one or more cesarean sections
* Gestational age: > 32 weeks
* The following ultrasound markers such as "loss of clear retroplacental translucency", "myometrial thinning", "abnormal lacunae", "irregular bladder wall", "utero-vesicalhypervascularity".
* Preoperative hemoglobin more than 10 gm/dl
* Cases with PAS that will undergoing CS Hysterectomy

Exclusion Criteria:

* Maternal medical disorders e.g.: coagulation defects, cardiac diseases etc.….
* Any known or reported hypersensitivity to the used medication.
* All cases with spontaneous placental separation at laparotomy.
* All patients undergoing conservative management of PAS.
* All cases which necessitate emergency termination.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | during operation
  amount of intraoperative blood loss in patients with PAS disorders undergoing cesarean hysterectomy

SECONDARY OUTCOMES:
operative time | during operation

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt